CLINICAL TRIAL: NCT06093490
Title: A Mobile Health Application to Detect Absence Seizures Using Hyperventilation and Eye-Movement Recordings
Brief Title: Detecting Absence Seizures Using Hyperventilation and Eye Movement Recordings
Acronym: DASHER
Status: Completed | Type: Observational
Sponsor: Eysz, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Rachel Kuperman, Principal Investigator, Eysz, Inc.
Other Study IDs: 1R43NS129363 (NIH); 1R43NS129363 (NIH)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Absence Epilepsy, Childhood; Absence Seizures; Absence Epilepsy; Epilepsy in Children; Staring; Seizures
Keywords: absence seizures; absence epilepsy; hyperventilation; staring spells
MeSH Terms: conditions — Epilepsy, Absence; Seizures; Hyperventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Absence Seizure: Age 4-12, Typical Absence Seizure captured during hyperventilation
  Interventions: Device: Eysz Hyperventilation Recorder
- Control Group: Age 4-12, Control Group without seizure activity during hyperventilation
  Interventions: Device: Eysz Hyperventilation Recorder

INTERVENTIONS:
Device: Eysz Hyperventilation Recorder — App used to guide and record hyperventilation

SUMMARY:
This study is being done to find out if a smartphone app can identify absence seizures. Children who have a history of absence seizures, as well as children without any seizure history, will be testing out the app. If participating the child will be guided through hyperventilation, an activity that asks the child to take quick, deep breaths. The app will record video of the child's face and sounds they make during hyperventilation. Hyperventilation is a safe and established technique frequently used during EEG (electroencephalogram) to encourage seizure occurrence. The App will be used during a regularly scheduled EEG.

DETAILED DESCRIPTION:
This observational study focuses on validating the use of the Eysz mHealth App - a smartphone-based tool for guided Hyperventilation (HV) and data collection - to aid clinicians in identifying absence seizures in people at risk for childhood absence epilepsy (CAE). The Eysz mHealth app will guide users through HV via interactive graphics while capturing audio and video data using smartphone sensors (e.g., camera, microphone) from which eye movements, facial biometrics/ expressions, number and length of exhales will be extracted.

The goal of this observational study is to determine an epileptologist's performance in identifying HV-induced absence seizures using video data collected from a smartphone when compared to the gold standard interpretation of the EEG. The exploratory goal is to develop machine learning based algorithms to identify HV-induced seizures.

ELIGIBILITY:
Inclusion Criteria:

* typical absence seizure during use of the Eysz Hyperventilation Recorder or Control

Exclusion Criteria:

* Other seizure type besides typical absence seizure during use of the Eysz Hyperventilation Recorder
* subclinical seizure activity
* inability to participate with study procedures
* contraindications to hyperventilation including history of subarachnoid hemorrhage, sickle cell anemia, recent cerebrovascular accident or myocardial infarction, significant cardiopulmonary disease, active asthma, known aneurysm, known moyamoya disease, or pregnancy.
* People who have a history of generalized tonic clonic convulsions (GTCs) provoked by hyperventilation

Ages: 4 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children undergoing routine EEG as part of clinical care at risk or known to have childhood absence epilepsy who will be undergoing hyperventilation
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of Eysz Hyperventilation (HV) Recorder Compared to video EEG (VEEG) | epileptologist review of 5 minutes of use of the Eysz Hyperventilation Recorder
  Voluntary HV triggers seizures in >90% of people with absence epilepsy and is a standard clinical procedure to assist in diagnosing and monitoring absence epilepsy. Clinical studies have shown HV to be a safe and effective procedure. This study focuses demonstrating the accuracy of the physician read of a smartphone video generated by the Eysz Hyperventilation (HV) Recorder- a smartphone-based tool for guided HV and video data collection. Three epileptologists will review the VEEG during use of the Eysz HV Recorder to identify typical absence seizures. Three independent epileptologists will review the concurrently generated video from the Eysz HV Recorder to identify typical absence seizures.
  Our primary endpoint is that the lower bound of the 95% confidence interval of the accuracy of the majority classification of the smartphone video is ≥ 75% in comparison to the majority classification of the VEEG by 3 independent expert reviewers.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No